CLINICAL TRIAL: NCT01617330
Title: Controlled Exposure to Diesel Exhaust in Subjects With Allergic Rhinitis
Acronym: DALLER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Umeå (Other)
Collaborators: King's College London (Other)
Responsible Party: Principal Investigator, Dr Annelie F Behndig, MD PhD, MD PhD, University Hospital, Umeå
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: DALLER
Record Dates: First submitted 2012-06-05; First posted 2012-06-12 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Allergic Rhinitis
Keywords: Particulate matter; Air pollution; Diesel exhaust; Allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Bronchoscopy; Particulate Matter; Air Pollution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diesel exhaust (Experimental): 2 hour exposure to diesel exhaust at 100 microgram per cubic meter during intermittent exercise
  Interventions: Procedure: Bronchoscopy
- Filtered air exposure (Experimental): 2 hour exposure to filtered air during intermittent exercise
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy — Bronchoscopy with endobronchial biopsy sampling and bronchoalveolar lavage (BAL) 18 hours post exposure. Airway inflammation was assessed.
  Other Names: Particulate matter; Air pollution; BAL

SUMMARY:
Proximity to traffic, particularly to diesel-powered heavy-duty vehicles, has been associated with inducing and enhancing allergies in children and adults. To investigate the basis for this association, a controlled exposure of allergic rhinitics to diesel exhaust was performed at a dose known to be pro-inflammatory in healthy individuals.

The hypothesis was that airway inflammation would be augmented in allergic rhinitics following exposure to diesel exhaust at an environmentally pertinent particulate matter concentration.

Fourteen allergic rhinitics were exposed in a double-blinded, randomised trial to both diesel exhaust at 100 microgram/m3 PM10 (representing an aerosol of nanoparticulate combustion particles, mean diameter 80 nm) and filtered air for two hours on separate occasions. Bronchoscopy with endobronchial mucosal biopsies and airway lavage was performed 18 hours post-exposure, and samples were analysed for markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* History of seasonal allergic rhinitis requiring medical treatment only during the pollen season and were classified as mild and intermittent according to ARIA guidelines.
* Positive skin prick test to airborne allergens
* Normal lung function
* Negative Metacholine challenge

Exclusion Criteria:

* Current smoking or a previous history of smoking.
* Asthma
* Chest infection within six weeks prior to or during the study
* Current use of non-steroidal anti-inflammatory drugs
* Current vitamin C or E supplementation
* Current use of topical nasal steroids.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2001-03; Primary Completion 2002-02 (Actual); Study Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
Airway inflammation | 18 hours post exposure
  Bronchoscopy with endobronchial mucosal biopsies and airway lavage was performed 18 hours post-exposure to diesel exhaust and filtered air, and samples were analysed for markers of inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Annelie F Behndig, MD PhD, Principal Investigator — Department of Public Health and Clinical Medicine, Division of medicine, Umeå University, Umeå
Locations (1):
- Department of Public Health and Clinical Medicine, Division of medicine, Pulmonary medicine, Umeå, Sverige, Sweden

REFERENCES:
- [Background] Morgenstern V, Zutavern A, Cyrys J, Brockow I, Koletzko S, Kramer U, Behrendt H, Herbarth O, von Berg A, Bauer CP, Wichmann HE, Heinrich J; GINI Study Group; LISA Study Group. Atopic diseases, allergic sensitization, and exposure to traffic-related air pollution in children. Am J Respir Crit Care Med. 2008 Jun 15;177(12):1331-7. doi: 10.1164/rccm.200701-036OC. Epub 2008 Mar 12. PMID 18337595
- [Background] Gehring U, Wijga AH, Brauer M, Fischer P, de Jongste JC, Kerkhof M, Oldenwening M, Smit HA, Brunekreef B. Traffic-related air pollution and the development of asthma and allergies during the first 8 years of life. Am J Respir Crit Care Med. 2010 Mar 15;181(6):596-603. doi: 10.1164/rccm.200906-0858OC. Epub 2009 Dec 3. PMID 19965811
- [Background] Oftedal B, Brunekreef B, Nystad W, Nafstad P. Residential outdoor air pollution and allergen sensitization in schoolchildren in Oslo, Norway. Clin Exp Allergy. 2007 Nov;37(11):1632-40. doi: 10.1111/j.1365-2222.2007.02823.x. Epub 2007 Sep 17. PMID 17877765
- [Background] Behndig AF, Larsson N, Brown JL, Stenfors N, Helleday R, Duggan ST, Dove RE, Wilson SJ, Sandstrom T, Kelly FJ, Mudway IS, Blomberg A. Proinflammatory doses of diesel exhaust in healthy subjects fail to elicit equivalent or augmented airway inflammation in subjects with asthma. Thorax. 2011 Jan;66(1):12-9. doi: 10.1136/thx.2010.140053. Epub 2010 Sep 13. PMID 20837873
- [Result] Brown JL, Behndig AF, Sekerel BE, Pourazar J, Blomberg A, Kelly FJ, Sandstrom T, Frew AJ, Wilson SJ. Lower airways inflammation in allergic rhinitics: a comparison with asthmatics and normal controls. Clin Exp Allergy. 2007 May;37(5):688-95. doi: 10.1111/j.1365-2222.2007.02695.x. PMID 17456216